CLINICAL TRIAL: NCT04141735
Title: A Real-life Study About Prediction of Sinusoidal Obstruction Syndrome With Ultrasound and Elastography Before Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Detection of Sinusoidal Obstruction Syndrome With Ultrasound After Allogeneic HSCT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: SOS detection CHU Nancy
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Sinusoidal Obstruction Syndrome
Keywords: SOS
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients from September 2016 to September 2018: all patients underwent allogeneic hematopoietic stem cell transplantation
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — no intervention

SUMMARY:
We would like conduct a real-life study in our center to evaluate the early detection of sinusoidal obstruction syndrome with hepatic ultrasound or elastography before allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The diagnosis of sinusoidal obstruction syndrome also know as veno-occlusive disease is often difficult. This is a potentially life-threatening complication that can develop after allogeneic hematopoietic stem cell transplantation. Clinically, sinusoidal obstruction syndrome is charaterized by hepatomegaly, right upper quadrant pain, jaundice and ascites. The diagnosis is based on biological parameters (bilirubin increase ≥ 2mg/dL or 34.2µmol/L) and clinical evaluation (sodium fluid retention with weight gain > 5%, ascites, painful hepatomegaly) (reference : M. Mohty and al. Revised criteria for sinusoidal obstruction syndrome, Bone Marrow Transplantation (2016) 906-912).

Early therapeutic intervention is pivotal for survival in sinusoidal obstruction syndrome, thus a rapid and reliable diagnosis has to be made. To rule out major differential diagnosis, a reliable imaging method is needed. In practice, doppler ultrasonography, is helpful to detect hepatomegaly and ascites but also is an help to explore well defined criteria of sinusoidal obstruction syndrome already published. For sonography criteria: hepatomegaly (3 measures) with an increase of 2cm versus baseline, gallbladder wall thickening, ascites or 3 criteria of a native VOD; splenomegaly, increase of the portal vein diameter, decrease of the hepatic vein diameter, visualisation of the para umbilical vein and for the doppler : increase of the hepatic artery RI (>0.75), monophasic flow in the hepatic veins (venous retraction is very typical but very late), flow demodulation on portal vein, decrease in portal flow, portal flow congestion, reversed flow, flow recorded in the para-umbilical vein ; all five last signs are late (reference : Lassau N. et al Prognostic value of doppler ultrasonography in hepatic veno occlusive disease. Transplantation 2002 jul 15 ;74(1) :60-6). These criteria can confirm the diagnosis : 6 signs of wich the first 3 can affirm the diagnosis with certainty in combination with clinical and biological parameters. There is currently a few data in the literature about prediction or early detection of this complication with systematic ultrasound +/- elastography. In this study, we want to evaluate in a real-life study the interest of this technique in the early and systematic prediction/ detection of sinusoidal obstruction syndrome.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with allogeneic hematopoietic stem cell transplantation in Nancy University Hospital between Sep 2016 and dec 2024

Exclusion Criteria:

* age < 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients transplanted for hematologic disease
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
incidence in the cohort of sinusoidal obstruction syndrome | up to 24 months
  incidence

CONTACTS AND LOCATIONS:
Overall Officials: Maud D'Aveni, MD, PhD, Principal Investigator — Université de Lorraine - CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Dignan F, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Okamoto S, Pagliuca A, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Duarte RF, Carreras E. Revised diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in adult patients: a new classification from the European Society for Blood and Marrow Transplantation. Bone Marrow Transplant. 2016 Jul;51(7):906-12. doi: 10.1038/bmt.2016.130. Epub 2016 May 16. PMID 27183098
- [Background] Lassau N, Auperin A, Leclere J, Bennaceur A, Valteau-Couanet D, Hartmann O. Prognostic value of doppler-ultrasonography in hepatic veno-occlusive disease. Transplantation. 2002 Jul 15;74(1):60-6. doi: 10.1097/00007890-200207150-00011. PMID 12134100